CLINICAL TRIAL: NCT01676181
Title: Randomised Surgical Intervention Study Between Adenotonsillectomy and Adenotonsillotomy in Children With Obstructive Sleep Apnea Syndrome
Brief Title: ATT Compared With ATE in OSAS Children
Acronym: RCT ATE/ATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Danielle Friberg, Associate Professor, senior surgeon, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/333-31/4
Record Dates: First submitted 2012-08-21; First posted 2012-08-30 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea Syndrome in Children
Keywords: Obstructive sleep apnea syndrome; Children; Polysomnography; Surgery; Coblation; Tonsils; Tonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adenotonsillectomy (Active Comparator): Total removal of tonsils and adenoids with cold steel
  Interventions: Procedure: Adenotonsillectomy
- Adenotonsillotomy (Active Comparator): Partial removal of tonsils with coblation and total removal of adenoids with cold steel
  Interventions: Procedure: Adenotonsillotomy

INTERVENTIONS:
Procedure: Adenotonsillectomy — Total removal of tonsils and adenoid tissue with cold-steel
  Arms: Adenotonsillectomy
Procedure: Adenotonsillotomy — Partial removal of tonsils with coblation and total removal of adenoids with cold steel
  Arms: Adenotonsillotomy

SUMMARY:
Non-inferiority hypothesis; adenotonsillotomy is equally good as adenotonsillectomy in treating obstructive sleep apnea syndrome (OSAS) in children after one, three and ten years.

DETAILED DESCRIPTION:
Background: Children with obstructive sleep apnea syndrome (OSAS) have apneas and disturbed sleep, which causes daytime symptoms such as neurobehavioral problems. OSAS is a significant cause of morbidity among children with an incidence of 1-3%, and a peak prevalence at 2-5 years of age. If left untreated it can cause severe complications including failure to thrive, cardiovascular complications, metabolic conditions and neurobehavioral disturbances (eg hyperactivity, inattention).

Golden standard to diagnose OSA in children is full-night polysomnography (PSG) at a sleep laboratory including EEG, EOG, EMG, video-audiometry and respiratory recordings. At the Department of Otorhinolaryngology at Karolinska University Hospital, we have a sleep laboratory performing in-lab full-night polysomnography.

The cause of OSAS in children is usually adenotonsillar hypertrophy, and the treatment of choice is surgical removal of tonsils and adenoid. Traditionally total adenotonsillectomy (ATE) has been performed, but in the last decade an alternative surgical method with partial adenotonsillotomy (ATT) is developed, where only the medial portion of the tonsil is removed. The newer method ATT is not fully evaluated in comparison with traditional ATE. There are studies comparing evaluating post-operative pain and bleeding showing a slight advantage for the TT-method. Very few studies are performed using objectively measured PSG-parameters to evaluate the effect of surgery on the sleep fragmentation and the sleep apneas. There is a need for such studies in the field of surgical treatment of pediatric OSA. This was also stated in a Cochrane database review from 2009, in which the conclusion was that there is a need for high quality randomised controlled trials to be carried out investigating the efficacy of surgical treatment of OSA in children. This makes this study important and of high clinical interest.

Aims: To increase the knowledge of pediatric OSA and its treatment and to optimize the surgical treatment for children with OSA.

To through a blinded randomized controlled trial compare the efficacy of ATT and ATE in treating OSA in children, including long-term follow-up after one, three and ten years.

To evaluate postoperative pain after ATE and ATT. To evaluate quality of life after ATE and ATT.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-6 years
* Clinical symptoms of OSAS (apneas, snoring, disturbed sleep)
* Tonsil size 3-4 with the Brodsky scale (obstructing at least 50% of the oro-pharyngeal space)
* Apnea-Hypopnea Index (AHI) 5-30 (moderate- severe OSA)

Exclusion Criteria:

* Clinical signs of craniofacial anomalies or neuromuscular disorders
* Obesity
* Earlier having had surgery of tonsils or adenoid
* Bleeding disorder
* Cardiopulmonary disorder

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2011-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in polysomnographic parameter AHI (Apnea Hypopnea Index) | One, three and ten years
  AHI; the number of apneas and hypopneas per sleep hour, is measured through polysomnography before and after surgery.

SECONDARY OUTCOMES:
Changes in quality of life questionnaires (OSA18 and SDQ) | One, three and ten Years
  Parents answering to quality of life-questionnaire OSA18 and SDQ (Strengths and Difficulties Questionnaire) before and after surgical intervention

OTHER OUTCOMES:
Per- and postoperative bleeding | One year
  The two groups (ATT and ATE) will be compared concerning per- and postoperative bleeding.
changes in polysomnographic parameters other than AHI | one, three and ten years
  Polysomnograhic parameters, for example; the oxygen desaturation index (ODI), lowest oxygen saturation, the respiratory disturbance index (RDI), AHI in REM, total sleep time, time in REM, deep sleep, supine position etc.
Differences in postoperative pain | One year
  The two groups will be compared with questionnaires and consumption of analgetics concerning the degree of postoperative pain.
Number of patients who need reoperations | One, three and ten years
  The patient may need reoperations, either because of postoperative bleeding or because the tonsils have regrowth
Abnormalities in DNA analysis of blood and tonsil tissue | one year
  Blood and tissue samples will be frozen for future analysis of DNA. We have not yet decided which method we will use. There are other studies suggesting abnormalities in certain enzymes in children with tonsillar hypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friberg, MD, PhD, Principal Investigator — Karolinska University Hospital, ORL dep
Locations (1):
- Karolinska University Hospital, ORL dep, Stockholm, Sweden

REFERENCES:
- [Derived] Blackshaw H, Springford LR, Zhang LY, Wang B, Venekamp RP, Schilder AG. Tonsillectomy versus tonsillotomy for obstructive sleep-disordered breathing in children. Cochrane Database Syst Rev. 2020 Apr 29;4(4):CD011365. doi: 10.1002/14651858.CD011365.pub2. PMID 32347984
- [Derived] Borgstrom A, Nerfeldt P, Friberg D. Postoperative pain and bleeding after adenotonsillectomy versus adenotonsillotomy in pediatric obstructive sleep apnea: an RCT. Eur Arch Otorhinolaryngol. 2019 Nov;276(11):3231-3238. doi: 10.1007/s00405-019-05571-w. Epub 2019 Aug 3. PMID 31377901